CLINICAL TRIAL: NCT00955526
Title: Placebo-Controlled, Double-Blind, Parallel Group, Fixed Dose Study of KW-6002 (Istradefylline) in the Treatment of Parkinson's Disease (Phase 3)
Brief Title: Study of KW-6002 (Istradefylline) for the Treatment of Parkinson's Disease in Patients Taking Levodopa
Acronym: 6002-009
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-009
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; levodopa; end of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Istradefylline 20mg (Experimental)
  Interventions: Drug: Istradefylline
- Istradefylline 40mg (Experimental)
  Interventions: Drug: Istradefylline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Istradefylline — 20 mg KW-6002 per day (two 10 mg tablets orally once daily for 12 weeks)
  Other Names: KW-6002
  Arms: Istradefylline 20mg
Drug: Istradefylline — 40mg KW-6002 per day (two 20 mg tablets orally once daily for 12 weeks)
  Other Names: KW-6002
  Arms: Istradefylline 40mg
Drug: Placebo — Two placebo tablets once daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish the efficacy of 20 mg/day and 40 mg/day doses of istradefylline for reducing the mean total hours of awake time per day spent in the OFF state in patients with advanced Parkinson's disease (PD) treated with levodopa. Patients who meet entry criteria will be randomized in a 1:1:1 ratio to double blind treatment with oral doses of 20 or 40 mg/day istradefylline or matching placebo. Patients will be treated for 12 weeks and will have interim visits and end of treatment visit to assess the efficacy and safety of istradefylline.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to give written informed consent
2. UK Parkinson's Disease Society (UKPDS) brain bank criteria (Step 1 and 2) for PD
3. PD stages 2-4 in the OFF state for Modified Hoehn and Yahr Scale
4. On levodopa/dopa-decarboxylase inhibitor for at least one year
5. Taking at least three doses and >=300 mg of levodopa/dopa-decarboxylase inhibitor per day for at least four weeks before randomization
6. Predictable end of dose wearing off
7. Able to satisfactorily complete Hauser based 24-hour patient Parkinson's diary
8. Have an average of two hours of OFF time on 24-hour diaries
9. On a stable regimen of any other anti-Parkinson's drugs for at least four weeks before randomization
10. On a stable dose of domperidone for at least 14 days before randomization

Exclusion Criteria:

1. Taking any excluded medications
2. Neurosurgical treatment or Transcranial Magnetic Stimulation for PD
3. Diagnosis of cancer within 5 years
4. Diagnosis of clinically significant illness of any organ system
5. Diagnosis of dementia or mini-mental status examination score of 23 or less
6. History of drug or alcohol abuse or dependence within the past two years
7. History of psychosis
8. History of significant drug allergies
9. Taking anticonvulsants for seizures
10. History of neuroleptic malignant syndrome
11. Pregnant or lactating females

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Reducing the mean total hours of awake time per day spent in the OFF state

SECONDARY OUTCOMES:
Reducing the mean percentage of awake time per day spent in the OFF state
Mean change in the total hours and the percentage of awake time per day spent in the ON state (without dyskinesia, with dyskinesia, with non-troublesome dyskinesia, and with troublesome dyskinesia)
Change in Unified Parkinson's Disease Rating Scale (UPDRS)
Change in the Clinical Global Impression - Improvement scale (CGI-I)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Tokyo, Japan